CLINICAL TRIAL: NCT01394406
Title: Effect of Ketamine Added to Intravenous Patient-controlled Analgesia on Postoperative Pain, Nausea and Vomiting in Patients Undergoing Lumbar Spinal Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 4-2009-0670
Record Dates: First submitted 2011-07-13; First posted 2011-07-14 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-03

CONDITIONS: Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Ketamine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ketamine group (Experimental)
  Interventions: Drug: Ketamine
- Saline group (Placebo Comparator)
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Ketamine — ketamine 3 mg/kg mixed to intravenous patient controlled analgesia device (fentanyl 20 mcg/kg. total volume 180 ml, basal infusion 2 ml, bolus 2ml, lock-out 15 min)
  Arms: Ketamine group
Drug: Saline — equal volume of normal saline mixed to intravenous patient controlled analgesia device
  Arms: Saline group

SUMMARY:
Ketamine added to intravenous patient-controlled analgesia may be effective on prevention of postoperative nausea and vomiting by reducing opioid requirement after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking female patients undergoing elective lumbar spinal surgery
* Age 20-65
* American Society of Anesthesiologists physical status classification I or II

Exclusion Criteria:

* Antiemetic within 24 hrs, Taking Steroids, Opioids within 1 week
* Psychiatric disease, Active drug or alcohol abuse
* GI motility disorder, severe renal/ hepatic disease
* insulin-dependent DM
* admission to ICU after surgery

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-01; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative nausea and vomiting | within 48 hrs after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea